CLINICAL TRIAL: NCT03733340
Title: Antibacterial Prophylaxis With Imipenem vs no Prophylaxis for Hematological Malignancies Patients Before Allogenetic Hematopoietic Stem Cell Transplantation
Brief Title: Antibacterial Prophylaxis vs no Prophylaxis for Hematological Malignancies Patients Before Allo-HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Prof., Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Bacteria clean pre-allo-HSCT
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-08

CONDITIONS: Antibacterial Prophylaxis; Hematological Malignancies; Allogenetic Hematopoietic Stem Cell Transplantation; Imipenem
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Imipenem

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imipenem prophylaxis group (Experimental): Imipenem: 1g q8h i.v. daily for 5 consecutive days before the onset of conditioning of allo-HSCT
  Interventions: Drug: Imipenem
- Blank control group (No Intervention): Without antibacterial prophylaxis at the onset of condition of all-HSCT

INTERVENTIONS:
Drug: Imipenem — Imipenem: A wide-spectre antibiotic from the carbapenem group Other name: Imipenem-cilastatin
  Arms: Imipenem prophylaxis group

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is a potentially curative treatment for a variety of hematologic malignancies. Bacterial infections remain a common complication of allo-HSCT, especially in the pre-engraftment phase. Pre-engraftment neutropenia typically lasts for up to 2 weeks in autologous HSCT but is considerably longer in allogeneic HSCT recipients who receive myeloablative conditioning regimens. This is a prospective, randomized, controlled, phase II/III clinical trial that aims to investigate the beneficial and harmful effects of prophylactic use of imipenem in patients with hematological malignancies before allo-HSCT. All patients aged above 14 years, diagnosed with hematological malignancies and ready to undergo allo-HSCT, no active infection within 3 weeks before allo-HSCT, with a normal CT scan-chest before entering the transplantation cabin and willing to participate in the trial will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* aged above 14 years;
* diagnosis with hematological malignancies and be ready to undergo allo-HSCT;
* no active infection within 3 weeks before allo-HSCT;
* with a normal CT scan-chest before entering the transplantation cabin.

Exclusion Criteria:

* age < 14 years;
* active and documented infection at admission;
* with a abnormal CT scan-chest before entering the transplantation cabin;
* with any conditions not suitable for the trial;
* unwilling to participate in the trial.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Infectious incidence | pre-engraftment in allo-HSCT

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
Incidence of acute GVHD | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Liu Qifa, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided